CLINICAL TRIAL: NCT07048808
Title: Endocardial Delivery of XC001 Gene Therapy for Refractory Angina Coronary Treatment: A 26-Week (With 26 Week Extension) Phase 2b Randomized, Multi-Center, Double-Blind, Sham Controlled Study to Evaluate Efficacy and Safety
Brief Title: Investigational Trial to Evaluate XC001 Delivered Via an Cardiac Catheter in Subjects With Chronic Angina.
Acronym: EXACT2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: XyloCor Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XC001-1002
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Refractory Angina; Coronary Artery Disease
Keywords: Angina; EXACT 2; Refractory angina
MeSH Terms: conditions — Angina Pectoris; Coronary Artery Disease | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, sham-procedure control study. Subjects with RA (CCS class II-IV) with no therapeutic options will be randomized 1:1 to either the treatment group with catheter delivery of 4×1011 vp XC001 (approximately N=53) or a sham procedure group (approximately N=53).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded trial, there is a blinded team at the CRO
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Active Comparator): Those randomized to the treatment group will have XC001 administered by percutaneous catheter delivery using the Extroducer® Infusion Catheter System (delivery catheter).
  Interventions: Combination Product: XC001
- Sham group (Sham Comparator): Subjects randomized to the sham catheterization procedure group will receive the same procedure as the treatment group (with introduction of an iliofemoral or radial sheath, positioning of the pigtail catheter in the left ventricle, generation of ventriculograms, and mimicking of the injection procedure by the interventional team following a Cath Lab script), except they will not have the delivery catheter inserted and will not receive any endocardial injections
  Interventions: Combination Product: Sham (No Treatment)

INTERVENTIONS:
Combination Product: XC001 — XC001 administered by percutaneous catheter delivery using the Extroducer® Infusion Catheter System.
  Arms: Treatment group
Combination Product: Sham (No Treatment) — Subjects randomized to the sham catheterization procedure group will receive the same procedure as the treatment group (with introduction of an iliofemoral or radial sheath, positioning of the pigtail catheter in the left ventricle, generation of ventriculograms, and mimicking of the injection procedure by the interventional team following a Cath Lab script), except they will not have the delivery catheter inserted and will not receive any endocardial injections
  Arms: Sham group

SUMMARY:
This is a two-part study, comprised of an initial open-label run-in phase (Part 1) in a subset of 3 subjects to provide first data regarding safety, and feasibility of the percutaneous endovascular catheter-facilitated intramyocardial delivery of XC001 in patients with RA due to obstructive CAD.

Part 1 of the study is comprised of 3 subjects with RA (CCS class II-IV) who will receive 4×1011 viral particles (vp) XC001. An Independent Data Monitoring Committee (IDMC), the committee will review safety and feasibility data and approval to commence enrollment in Part 2 of the study.

Part 2 is a randomized, double-blind, sham-procedure control study. Subjects with RA (CCS class II-IV) with no therapeutic options will be randomized 1:1 to either the treatment group with catheter delivery of 4×1011 vp XC001 (approximately N=53) or a sham procedure group (approximately N=53). It is estimated that approximately 106 subjects will be randomized to result in 100 evaluable subjects. All subjects enrolled in Part 1, as well as Part 2 will follow all screening and safety monitoring procedures for up to 12 months (Table 2), and will be included in the safety analysis of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age 18 to 85 years, inclusive, at the time of signing the ICF.
2. Diagnosis of chronic angina due to obstructive CAD that is refractory to drug therapy and unsuitable for revascularization via coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI) (as defined by ESC Joint Study Group on the Treatment of Refractory Angina Refractory, Mannheimer et al, EHJ 2002 and the 2013 ESC guidelines on the management of stable coronary artery disease, Montalescot et al, EHJ 2013; and Jolicoeur et al 2008).
3. Angina class II-IV as measured by CCS Functional Classification of Angina Pectoris.
4. History of evidence of reversible left ventricular ischemia, as assessed by stress ECG (including screening), stress echocardiography, single- photon emission computed tomography (SPECT), CT angiography imaging with fractional flow reserve analysis, stress PET (including screening) or cardiac magnetic resonance (CMR) imaging that has not resolved with intervention or by an acute coronary event.
5. Coronary angiography (and/or computed tomography (coronary) angiography (CTA)) within the past 18 months unless there is a clinical indication to warrant a more current procedure as determined by the investigator.
6. Two baseline ECG stress tests (treadmill test, modified Bruce protocol) that adhere to the following (details outlined in the ETT manual):

   i. A modified Bruce protocol that includes two three-minute warm- up stages of 1.7 mph/ 0% grade and 1.7 mph/ 5% grade.

   ii. TED of 90 seconds to 9.5 minutes that is limited/stopped because of angina (or angina equivalent).

   iii. The maximally allowed variation between two subsequent treadmill tests should not exceed 25% and should not exceed 75 seconds. The ETT core laboratory must review and approve the ETTs for eligibility.

   iv. The tests must be performed at least 48 hours apart from each other. v. A third test is permitted if the second test does not meet the criteria.
7. On a stable regimen of anti-anginal, anti-hypertensive, and lipid lowering medications deemed medically appropriate for RA at the discretion of the investigator. The chronic anti-anginal regimen must include at least two functional classes at the maximally tolerated dose for the preceding 30 days prior to the screening visit (Jolicoeur 2008). Functional classes include beta-blockers, calcium channel blockers, (long-acting) nitrates, and metabolic modulators (i.e., ranolazine, trimetazidine, ivabradine, nicorandil). Use of fewer than two functional classes may be allowed if there is evidence of intolerance to those classes of anti-anginal medications.
8. Formally approved by the ERC to undergo the study procedure by a review of past medical history and screening assessments, with emphasis on reversible left ventricular ischemia (further details provided in the ERC Charter).
9. All subjects capable of procreation with their partners must agree to use a highly effective and medically accepted method of contraception for 6 months following the study procedure (Day 1) to avoid pregnancy (as defined in Appendix A). This is not required of female subjects who are either:

   * Postmenopausal (defined as no menses for 12 months without an alternative medical cause) prior to screening. In addition, at least 2 high follicle stimulating hormone (FSH) measurements in the postmenopausal range must be used to confirm a postmenopausal state in women with less than 12 months of amenorrhea and not using hormonal contraception or hormonal replacement therapy; OR
   * Surgically sterile (i.e., hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) at least 1 month prior to Screening
10. Female subjects agree to not donate oocytes and male subjects must agree not to donate sperm for 6 months following administration of the investigational product (IP).
11. Capable of providing informed consent and undergoing all the required tests and procedures in the protocol.

Exclusion Criteria:

1. Any of the following:

   1. ST-Elevation or non-ST elevation myocardial infarction (STEMI or NSTEMI) not requiring revascularization, transmural MI, or cerebral vascular accident within the past 60 days prior to the screening visit.
   2. Uncontrolled hypercholesterolemia defined as low-density lipoprotein (LDL) above 190 mg/dL.
   3. Uncontrolled hypertension (systolic blood pressure [BP] >180 mmHg, diastolic BP >100 mmHg) despite maximal medical treatment.
   4. Current untreated malignant ventricular arrhythmias (with episode of sustained or non-sustained ventricular tachycardia (VT) in last 30 days; suspected/probable/definite).
   5. Current untreated bradyarrhythmia (<50 bpm) for which a new artificial pacemaker placement is anticipated during the study period. A current pacemaker is allowed.
   6. Congestive heart failure defined as New York Heart Association Function Class III or IV or left ventricular ejection fraction < 25% within the 6 weeks prior to the screening visit (or as assessed by the screening contrast Echo).
   7. Anginal episodes that routinely require the administration of opiates.
2. Moderate to severe aortic valve stenosis (defined as Doppler echocardiography determined peak pressure gradient that exceeds 40 mm Hg (or Vmax >3.2 m/s) and/or subjects with a mechanical valve in the aorta valve position.
3. Presence of a ventricular thrombus (as defined by contrast transthoracic echocardiography at screening). Subjects may be rescreened after 6 weeks of adequate treatment and absence of ventricular thrombus by echocardiography.
4. Body mass index > 45 kg/m2.
5. Hemoglobin < 10 g/dL, absolute neutrophil count < 1.2 × 103 per µL, platelet count < 75,000 per µL, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 3 x upper limit of normal (ULN), total bilirubin > 2 x ULN unless the subject has a previously known history of Gilbert's syndrome and estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2
6. Diabetic with current glycosylated hemoglobin (HbA1c) > 9.5% or active proliferative diabetic retinopathy.
7. Documented active proliferative retinopathy from any cause (ETDRS [Early Treatment Diabetic Retinopathy Study] score >35).
8. Uncontrolled coagulation disorder (that cannot be corrected by pharmacotherapy)
9. Patients with unstable chronic obstructive pulmonary disease despite adequate treatment.
10. A history or evidence of human immunodeficiency virus (HIV) or active hepatitis C virus (HCV), or active hepatitis B virus (HBV).
11. Severely immuno-compromised patients, including high-dose chronic corticosteroid therapy or cytostatic (oncolytic) therapy.
12. Diagnosis of, or treatment for, any cancer within the last 5 years except for cutaneous basal or squamous cell carcinoma or carcinomas in situ where surgical excision was considered curative. (Past medical history of cancer is not exclusionary if the subject has been disease free for at least 5 years since the end of treatment).
13. Known hypersensitivity or any other contraindication to adenosine, regadenoson, or contrast agents used in any of the radiographic procedures or contraindication to anesthesia employed for the study procedure.
14. Pregnancy or currently lactating.
15. Receiving an investigational intervention or participating in another clinical trial within 30 days or within 5 half-lives of the drug prior to screening. Exception may be made if the individual is enrolled in a non- therapeutic observational study (registry) or the observational portion of a therapeutic study where the sponsoring authority authorizes enrollment.
16. Prior participation in any gene therapy; however, if the study was unblinded or documentation otherwise exists that the subject was randomized to the placebo control group and did not receive active gene transfer agent, the subject may be considered for this study. Has a serious or unstable medical or psychological condition (including drug or alcohol abuse) or other circumstance that, in the opinion of the investigator or ERC, would compromise the subject's safety or successful participation in the study or interpretation of study results. In particular, any suspected drug-seeking behavior related to chest pain should be exclusionary.
17. Known allergy to nickel.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint | 6 months
  The primary objective of this study is to evaluate the effect of XC001 on a composite endpoint of a) TED from a graded treadmill test (ETT), as assessed by a core lab, b) angina frequency from a diary (extracting the 2 weeks prior to the Week 12 and Week 26 visit) and c) ischemic burden, as quantified by stress imaging by PET (as assessed by a core lab) at 12 and 26 weeks following a one-time endocardial administration to CAD patients with RA compared to the sham procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Henry, MD, Principal Investigator — Christ Hospital
Locations (1):
- Christ Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No